CLINICAL TRIAL: NCT02184091
Title: An Open-Label, Single Dose Study to Evaluate the Effects of Underlying Renal or Hepatic Dysfunction on the Pharmacokinetics of Nevirapine (VIRAMUNE®)
Brief Title: Study to Evaluate the Effects of Underlying Renal or Hepatic Dysfunction on the Pharmacokinetics of Nevirapine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1259
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Renal Insufficiency; Hepatic Insufficiency
MeSH Terms: conditions — Renal Insufficiency; Hepatic Insufficiency | interventions — Nevirapine

ARMS (1):
- Nevirapine (Experimental): Single dose administration
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
Study to assess the effects of varying degrees of renal dysfunction and hepatic insufficiency on the single-dose pharmacokinetics of nevirapine and nevirapine metabolites in order to establish an appropriate dose and/or dosing frequency for renally- and hepatically-impaired patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any race between the ages of 18 and 75 years with weight within 30% of normal for gender, height and frame as specified by the Metropolitan Life Insurance Table
* For patients in the renal group: stable creatinine clearance based on two estimations taken at least 3 days apart, corresponding to one of four groups:

  * Group 1 (mild dysfunction) = 50 ml/min <= Creatinine Clearance (CLcr) < 80 ml/min
  * Group 2 (moderate dysfunction) = 30 ml/min <= CLcr < 50 ml/min
  * Group 3 (severe dysfunction) = CLcr < 30 ml/min and
  * Group 4 = end-stage renal disease (ESRD) requiring dialysis
* For patients in the hepatic group

  * Two baseline creatinine clearances (taken at least 3 days apart) > 80 ml/min
  * clinically diagnosed with hepatic insufficiency and Class A or B liver disease according to Child-Pugh's Classification; subjects must have a Child-Pugh score of 5-9 points
* For patients in the normal group, i.e. normal with respect to hepatic and renal function

  * matched with hepatic group regarding gender, age (+- 10 years), weight (+- 30 pounds) and smoking history
  * Two baseline creatinine clearances (taken at least 3 days apart) > 80 ml/min
  * No abnormalities on clinical or laboratory evaluations
* Female patients of childbearing potential must be willing to use a reliable form of contraception which must include a medically approved form of barrier contraception
* Patients who are able to provide written consent and comply with study requirements

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Seated systolic blood pressure either < 100 mmHg or > 150 mmHg and/or heart rate either < 50 beats/min or > 90 beats/min
* History of any illness or drug allergy that in the opinion of the investigator might confound the results of the study or pose additional risk in administering nevirapine to the subject
* Patients who have had an acute illness or hospitalization other than for routine dialysis within 2 weeks prior to study initiation
* Patients who are currently taking any over-the-counter drug within 3 days prior to study initiation, or who are currently taking any prescription drug that in the opinion of the investigator in consultation with Boehringer Ingelheim Pharmaceuticals Incorporated (BIPI) medical monitor and pharmacokineticist might interfere with the absorption, distribution or metabolism on the test drug
* Significant electrocardiogram (ECG) abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-01; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
AUC (Area under the plasma concentration time curve) | up to 7 days
Cmax (Maximum observed concentration of the analyte in plasma) | up to 7 days
Tmax (Time of maximum concentration of the analyte in plasma) | up to 7 days
T1/2 (Terminal half-life of the analyte in plasma) | up to 7 days
Vss/F (Volume of Distribution) | up to 7 days
MRT (Mean residence time of the analyte) | up to 7 days
CL/F (Apparent clearance of the analyte in plasma) | up to 7 days

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 21 days
Number of patients with abnormal changes in laboratory parameters | Screening, Day 0, Day 7